CLINICAL TRIAL: NCT04218890
Title: Urinary Tissue Factor (TF), Tissue Factor Pathway Inhibitor (TFPI) and Plasmin as Bio-markers in Early Diagnosis of Lupus Nephritis
Brief Title: TF, TFPI and Plasmin as Novel Bio-markers in Early Diagnosis of Lupus Nephritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayat salah, principal investigator, Assiut University
Other Study IDs: ASA2
Record Dates: First submitted 2019-12-28; First posted 2020-01-06 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SLE patients without lupus nephritis: 40 SLE patients
  40SLE patients( All SLE pt. satisfied the ACR criteria for SLE diagnosis) these patients will be without any evidences of nephritis
  Interventions: Diagnostic Test: Urinary tissue factor (TF), tissue factor pathway inhibitor (TFPI) and plasmin
- SLE patients with lupus nephritis: 40SLE patients with evidences of nephritis
  Interventions: Diagnostic Test: Urinary tissue factor (TF), tissue factor pathway inhibitor (TFPI) and plasmin
- healthy control group: 20 healthy subjects matched age and sex with be enrolled as healthy control group
  Interventions: Diagnostic Test: Urinary tissue factor (TF), tissue factor pathway inhibitor (TFPI) and plasmin

INTERVENTIONS:
Diagnostic Test: Urinary tissue factor (TF), tissue factor pathway inhibitor (TFPI) and plasmin — urinary sample

SUMMARY:
Urinary levels of plasmin ,TF , and TFPI are all elevated in active LN patients compared to inactive LN patients and healthy controls. All four proteins correlated with systemic disease activity and renal disease activity. Importantly, urine plasmin performed best among the four proteins in discriminating active LN from inactive disease, even better than traditional markers, such as anti ds DNA and complement C3. Furthermore, the combination of urine plasmin and TFPI showed higher specificity and negative predictive values than urine plasmin when compared to anti-ds DNA and complement C3

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a systemic autoimmune disease affects various organs, characterized by diverse autoantibodies production,mainly anti-DNA and anti-nuclear antibodies . It demonstrates variations in incidence,prevalence, disease activity and prognosis according to race and ethnicity . Lupus nephritis (LN) is one of the most frequent and severe clinical manifestations of SLE, it affects over 60% of SLE patients representing a leading cause of morbidity and mortality . Early diagnosis and monitoring of the disease flares are still challenging , although of the novel immunosuppressive drugs and biologics, which brought improvements in recent SLE/LN survival rates .

The American College of Rheumatology (ACR) guidelines for the treatment of lupus nephritis , recommend change in treatment if response to therapy has not been achieved after 6 months of induction therapy. However, response to therapy is not well defined. In addition, renal damage can occur within 6 months while waiting to define this response. Decision support tools could help define response at the start of induction therapy and have the potential to improve outcomes .

Use of laboratory parameters for LN such as creatinine clearance, anti-ds DNA, proteinuria, urine protein-to-creatinine ratio (U-PCR),and complement levels are undesirable. These markers are of less sensitivity and specificity for evolve renal activity and injury in LN.They are not directly correlated with kidney damage, which can arise before kidney function affection. Outbreak of nephritis may occur in any condition in absence and new rise in the level of proteinuria.

Kidney biopsy is a gold standard to assess the histological category of LN and the level of activity and chronicity in glomeruli. But, it is an invasive procedure and continual biopsies are inappropriate in the observing and follow up of LN . It may have sampling error because of extent number of glomeruli obtained for LN activity and chronicity. So , many studies are focusing on identifying non-invasive biomarkers for the early diagnosis and follow up of the disease and the therapy response.

Urine is easily collected and can reflect the underlying renal affection more accurately than serum. Therefore, urine bio-markers represent promising candidates for the early disease diagnosis and monitoring .Thus, novel urinary bio-markers, which are able to distinguish lupus kidney activity and its extremity, anticipate kidney outbreak, and observe treatment reciprocation and illness breakthrough are clearly obligatory . Urinary bio-markers are more sensitive for lupus nephritis;they can appear in urine before functional derangement .

Coagulation system disorders and hyper-coagulability state have been reported in lupus nephritis, also the frequency of thrombotic events was documented to be higher in SLE patients than in the general population, and these events were associated with poor outcome .Both thrombo-genic and thrombolytic cascades appear to be up-regulated in lupus nephritis, with proteins from both cascades appearing in the urine .

Urinary levels of plasmin ,TF and TFPI are all elevated in active LN patients compared to inactive LN patients and healthy controls. All four proteins correlated with systemic disease activity and renal disease activity. Importantly, urine plasmin performed best among the four proteins in discriminating active LN from inactive disease, even better than traditional markers, such as anti dsDNA and complement C3. Furthermore, the combination of urine plasmin and TFPI showed higher specificity and negative predictive values than urine plasmin when compared to anti-dsDNA and complement C3.

ELIGIBILITY:
Inclusion Criteria:

1. age >15 years
2. SLE patients fullfiling ACR diagnostic criteria

Exclusion Criteria:

1. Renal artery stenosis, congenital renal diseases ,renal tumor,other causes of GN
2. Pregnancy.
3. coagulation disorders
4. DM,HTN and the other connective tissue disease
5. Obesity
6. CKD

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Clinical data will be gathered and SLEDAI will be calculated based on chart review .SLE patients will then classified as having either active LN (ALN) or inactive LN (ILN). Active LN is defined as active urine sediment or proteinuria (rSLEDAI > 0). Inactive LN is defined as inactive urine sediment and no proteinuria (rSLEDAI = 0).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
The diagnostic utility of tissue factor ,, tissue factor pathway inhibitor and plasmin as biomarkers for early detection of lupus nephritis (LN) | 2023
  Urinay sample of 100 subjects (80 with SLE ,40 of them with LN,and 20 are healthy persons)will be collected as a morning sample& using ELISA test to detect the level of these bio-markers in the urine of these subjects
the correlation of these bio-markers to the clinical staging , the disease activity index and revised treatment . | 2023
  correlate the level of the markers with the renal biopsy staging and activity index using (International Society of Nephrology /Renal Pathology Society classification (ISN/RPS), and disease Activity Index (SLEDAI-2K & r SLEDAI)).

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Qin L, Stanley S, Ding H, Zhang T, Truong VTT, Celhar T, Fairhurst AM, Pedroza C, Petri M, Saxena R, Mohan C. Urinary pro-thrombotic, anti-thrombotic, and fibrinolytic molecules as biomarkers of lupus nephritis. Arthritis Res Ther. 2019 Jul 18;21(1):176. doi: 10.1186/s13075-019-1959-y. PMID 31319876
- [Background] Frijns R, Fijnheer R, Schiel A, Donders R, Sixma J, Derksen R. Persistent increase in plasma thrombomodulin in patients with a history of lupus nephritis: endothelial cell activation markers. J Rheumatol. 2001 Mar;28(3):514-9. PMID 11296951
- [Background] Ding H, Kharboutli M, Saxena R, Wu T. Insulin-like growth factor binding protein-2 as a novel biomarker for disease activity and renal pathology changes in lupus nephritis. Clin Exp Immunol. 2016 Apr;184(1):11-8. doi: 10.1111/cei.12743. Epub 2016 Jan 11. PMID 26616478
- [Background] Petri M, Kasitanon N, Lee SS, Link K, Magder L, Bae SC, Hanly JG, Isenberg DA, Nived O, Sturfelt G, van Vollenhoven R, Wallace DJ, Alarcon GS, Adu D, Avila-Casado C, Bernatsky SR, Bruce IN, Clarke AE, Contreras G, Fine DM, Gladman DD, Gordon C, Kalunian KC, Madaio MP, Rovin BH, Sanchez-Guerrero J, Steinsson K, Aranow C, Balow JE, Buyon JP, Ginzler EM, Khamashta MA, Urowitz MB, Dooley MA, Merrill JT, Ramsey-Goldman R, Font J, Tumlin J, Stoll T, Zoma A; Systemic Lupus International Collaborating Clinics. Systemic lupus international collaborating clinics renal activity/response exercise: development of a renal activity score and renal response index. Arthritis Rheum. 2008 Jun;58(6):1784-8. doi: 10.1002/art.23456. PMID 18512819